CLINICAL TRIAL: NCT01751477
Title: Oral Probiotics (Infloran®) for Prevention of Necrotizing Enterocolitis in Very Low Birth Weight Infants
Brief Title: Infloran® for Prevention of Necrotizing Enterocolitis
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Collaborators: Wilheminenspital der Stadt Wien (Unknown)
Responsible Party: Principal Investigator, Andreas Repa, MD, Medical University of Vienna
Other Study IDs: MUV-Neo3
Record Dates: First submitted 2012-12-14; First posted 2012-12-18 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Necrotizing Enterocolitis
Keywords: Very Low Birth Weight Infants; Probiotics; Necrotizing Enterocolitis
MeSH Terms: conditions — Enterocolitis, Necrotizing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Probiotics (Infloran): Very low birth weight Infants receiving 2 capsules/d Infloran starting in the first week of life
- Control: Very low birth weight Infants who did not receive Infloran (historical cohort)

SUMMARY:
Necrotizing enterocolitis (NEC) is one of the most devastating gastrointestinal emergencies in preterm neonates and a leading cause of death and morbidity.

The pathogenesis of NEC remains largely unclear, but it is widely considered as a multifactorial disease. Prematurity, enteral feeding, bacterial colonisation of the gut and intestinal ischemia have been proposed as major risk factors.

Probiotics may prevent NEC by improving the maturity and function of the gut mucosal barrier, modulating the immune system, promoting colonization of the gut with beneficial organisms and preventing colonization by pathogens.

A variety of clinical trials have evaluated the effect of different probiotic preparations on the occurrence of NEC in preterm infants. The results of recent metaanalyses suggest a benefit of probiotic bacteria in reducing the incidence of NEC and propose a change of practice.

The aim of the study is to evaluate the efficacy of the probiotic preparation Infloran® in reducing the incidence of NEC after implementation in clinical routine in preterm (< 34 weeks gestational age) very low birth weight infants compared to a historical cohort.

ELIGIBILITY:
Inclusion Criteria:

* Neonates admitted to the neonatal intensive care unit on day 1 of life
* Very low birth weight (<1500 gram)
* Prematurity < 34/0 weeks gestational age
* For group receiving probiotics: 230 infants born after the 20/Sep/2010 (i.e. date of introduction of Infloran in clinical routine)
* For control group (historical): 230 infants born before 2010

Exclusion Criteria:

* Malformation of the gut (omphalocele, gastroschisis, intestinal atresia)
* Death before seven days of life, except due to NEC
* Transfer to another hospital before 37 weeks of corrected gestational age, except those who were transferred to a partner clinic using the same protocol for probiotic supplementation
* For group receiving probiotics: Infants who did not receive Infloran® starting in the first week of life or stopped before 34 weeks gestational age, except infants who developed NEC (reason for discontinuation of Infloran)

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Very low birth weight Infants (<1500g birth weight)
Sampling Method: Probability Sample
Enrollment: 463 (Actual)
Dates: Start 2010-09; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Incidence of NEC | From birth to 37 weeks of gestational age (usually around 12 weeks)
  NEC stages 2 or 3 according to Bell´s modified staging of NEC

SECONDARY OUTCOMES:
Severity of NEC | From birth to 37 weeks of gestational age (usually around 12 weeks)
Influence of enteral feeding with human milk or formula on the incidence of NEC after the implementation of Infloran® | From birth to 37 weeks of gestational age (usually around 12 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Repa, MD, Principal Investigator — Medical University Vienna; Nadja Haiden, MD, Study Director — Medical University Vienna; Margarita Thanhäuser, MD, Study Chair — Medical University Vienna
Locations (2):
- Austria (2):
  - Medical University Vienna, Vienna
  - Wilheminenspital der Stadt Wien, Vienna

REFERENCES:
- [Result] Repa A, Thanhaeuser M, Endress D, Weber M, Kreissl A, Binder C, Berger A, Haiden N. Probiotics (Lactobacillus acidophilus and Bifidobacterium infantis) prevent NEC in VLBW infants fed breast milk but not formula [corrected]. Pediatr Res. 2015 Feb;77(2):381-8. doi: 10.1038/pr.2014.192. Epub 2014 Nov 25. PMID 25423074
- See also: Homepage Medical University Vienna — http://www.meduniwien.ac.at